CLINICAL TRIAL: NCT05458219
Title: A Phase 1a/b, Multicenter, Open-label, First-in-human Study of IBI343 in Subjects With Locally Advanced Unresectable or Metastatic Solid Tumors
Brief Title: A First-in-human Study of IBI343 in Subjects With Locally Advanced Unresectable or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Collaborators: Fortvita Biologics (USA)Inc. (Industry); TigerMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI343A101
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Unresectable or Metastatic Solid Tumors
MeSH Terms: interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3 arms (Experimental): Phase 1a Part 3: For monotherapy: 6 mg/kg Q3W was confirmed as the optimal dosing regimen for balancing clinical benefits and potential risks.
  In 1L G/GEJ AC and 1L PDAC cohort of the Phase Ia (Part 3) study, IBI343 combination therapy is proposed to be administered at doses of 4 mg/kg (Dose level 1) Q2W or 5 mg/kg (Dose level 2) Q2W in participants with G/GEJ AC and PDAC for the randomized study.
  Interventions: Drug: FOLFIRINOX/mFOLFIRINOX; Drug: mFOLFOX; Drug: IBI343
- Single arm (Experimental): Phase 1a Part 1 Dose Escalation: IBI343 will be administered intravenously (IV) at different dose levels following traditional 3+3 dose escalation design for following levels.
  Phase 1a Part 1 Dose Expansion: IBI343 will be administered at dose levels which is equal or lower than MTD. Each dose level contains no more than 30 subjects (including subjects in dose escalation) Phase 1a Part 2 Dose Optimization: IBI343 will be administered in parallel cohorts (randomized 1:1 ratio) to determine the optimal dose for the PDAC indication across China, Australia and the US (n=40). Dose levels 4.5mg/kg and 6mg/kg will be studied.
  Phase 1b Dose Extension: IBI343 will be administered at RP2D.
  Interventions: Drug: IBI343

INTERVENTIONS:
Drug: IBI343 — IBI343 will be administered intravenously (IV) on Day 1 of every 21-day cycle.
  Arms: Single arm
Drug: FOLFIRINOX/mFOLFIRINOX — FOLFIRINOX/mFOLFIRINOX will be administered IV Q2W on Days 1-3 every 2 weeks (14 days).
  Arms: 3 arms
Drug: mFOLFOX — mFOLFOX will be administered IV Q2W on Days 1-3 every 2 weeks (14 days) in each cycle after IBI343
  Arms: 3 arms
Drug: IBI343 — IBI343 will be administered IV Q2W on Day1 (14 days).
  Arms: 3 arms

SUMMARY:
This is a Phase Ia/Ib, multicenter, open-label, first-in-human study to evaluate the safety, tolerability, PK, and efficacy of IBI343 in participants with locally advanced unresectable or metastatic solid tumors. It is planned to be carried out in different countries or regions such as China, Australia and US.

There are three parts in phase Ia. Part 1 includes dose escalation and expansion phase and part 2 is designed for dose optimization for IBI343 monotherapy.

Part 3 1L G/GEJ AC and 1L PDAC cohorts will include an initial safety lead-in stage to confirm the tolerability of IBI343 in combination with chemotherapy in 1L PDAC and G/GEJ AC, followed by a randomized dose-optimization stage designed to further characterize safety, pharmacokinetics, and preliminary efficacy to inform selection of the recommended Phase 3 dose. Part 3 metabolite profiling cohort is designed to explore the payload metabolites in an advanced PDAC population.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria to be met for both Phase Ia and Phase Ib:

1. Has signed written Informed Consent Form (ICF), willing and able to comply with protocol-specified visits and related procedures.
2. Phase Ia dose escalation phase, Phase Ia part 3 metabolite profiling cohort，Phase Ia part 3 1L G/GEJ AC and 1L PDAC cohorts Safety Lead-in stage: Has at least 1 evaluable lesion according to RECIST v1.1; Phase Ia dose expansion and dose optimization phase, Phase Ia part 3 1L G/GEJ AC and 1L PDAC cohorts Dose optimization stage, Phase Ib: Has at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors RECIST v1.1.
3. Age ≥ 18 years, of either sex.
4. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
5. Has an expected survival ≥ 12 weeks.
6. Has adequate bone marrow and organ function. Defined as:

   • Hematology: ANC ≥ 1.5 × 109/L; Platelet count ≥ 100 × 109/L; Hemoglobin ≥ 9.0 g/dL, participants must not have received transfusion of blood products (including red blood cell suspension, apheresis platelets, cryoprecipitate, etc.), erythropoietin (EPO), G-colony stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF) within 7 days prior to blood sample collection;
   * Hepatic function: TBIL ≤ 1.5 × ULN (TBIL ≤ 3 × ULN is allowed for participants with Gilbert's syndrome); ALT and AST ≤ 2.5 × ULN for participants without liver metastasis and ≤ 5 × ULN for participants with liver metastasis; Albumin ≥ 28 g/L;
   * Renal function: estimated creatinine clearance ≥ 30mL/min (using Appendix 5. Calculation of Estimated Creatinine Clearance and Body Surface ).
   * Coagulation function: international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (participants receiving anticoagulant therapy with coagulation function within the above range are allowed).
7. Female participants of childbearing potential or male participants whose partners are female of childbearing potential are required to use effective contraceptive measures throughout the treatment period and for 6 months after the final treatment period.

Inclusion Criteria for Phase Ia Dose Escalation:

1. Participants with histopathologically confirmed unresectable locally advanced or metastatic malignant solid tumors that have failed or were intolerant to standard therapy or for whom no standard therapy is available.

Inclusion Criteria for Phase Ia Dose Expansion, Dose Optimization and Phase Ia Part 3 Metabolite Profiling Cohort:

1. Participants with histopathologically confirmed unresectable locally advanced or metastatic G/GEJ AC, PDAC, BTC, or other solid tumors (For Phase Ia Part 3 metabolite profiling cohort, only PDAC allowed) who have failed or were intolerant to standard therapy or for which no standard therapy is available.
2. * CLDN18.2-positive confirmed by pathological examination (in dose expansion phase, G/GEJ AC and PDAC preferentially enrolled *** moderate to high expression of CLDN18. 2; in dose optimization phase and Phase Ia Part 3 metabolite profiling cohort, G/GEJ AC preferentially enrolled **high expression of CLDN18.2 and PDAC preferentially enrolled ***moderate to high expression of CLDN18.2). For participants with previous anti-CLDN18.2 treatment (including but not limited to monoclonal antibodies, ADCs, CAR-T, etc.), tumor samples should be obtained post anti-CLDN18.2 therapy for CLDN18.2 expression evaluation.

Inclusion Criteria for Phase Ia Part 3 1L G/GEJ AC Cohort:

1. Participants with histopathologically confirmed unresectable locally advanced or metastatic G/GEJ AC who has not received previous systemic therapy. (For Safety Lead-in stage, participants who has received previous systemic therapy are permitted.) A prior (neo)adjuvant systemic therapy completed within 6 months prior to disease relapse or progression will be considered as having received previous systemic therapy.
2. Confirmed Her 2-negative (defined as IHC 0 or 1+, or IHC 2+ and negative by in situ hybridization) disease.
3. Confirmed combined positive score (CPS) <5 as determined by local IHC testing.
4. Participants must not have previously received topoisomerase inhibitor-based antibody-drug conjugate(s), unless given peri-operatively without evidence of resistance.
5. Participants must not have previously received anti-CLDN18.2 therapy.
6. *CLDN18.2-positive confirmed by pathological examination by central laboratory (For Dose optimization stage, G/GEJ AC enrolled participants with Claudin18.2 immunohistochemical membrane staining intensity 2+/3+ in ≥50% of tumor cells).

Inclusion Criteria for Phase Ia Part 3 1L PDAC Cohort:

1. Participants with histopathologically confirmed metastatic PDAC who has not received previous systemic therapy in the metastatic setting. (For Safety Lead-in stage, participants who has received previous systemic therapy are permitted.) A prior (neo)adjuvant systemic therapy completed within 12 months prior to disease relapse or progression will be considered as having received previous systemic therapy.
2. Participants must not have previously received anti-CLDN18.2 therapy.
3. Participants must not have previously received topoisomerase inhibitor-based antibody-drug conjugate(s), unless given peri-operatively without evidence of resistance.
4. *CLDN18.2-positive confirmed by pathological examination by central laboratory (For Dose optimization stage, PDAC enrolled # specified expression of CLDN 18.2)

Inclusion Criteria for Phase Ib Cohort A:

1. Histopathologically confirmed unresectable locally advanced or metastatic G/GEJ AC.
2. Have received at least 2 lines of systemic therapy [anti-PD-(L)1 + platinum, fluoropyrimidines, paclitaxel/docetaxel, or irinotecan; participants with HER2 overexpression (defined as 3 + or 2 + by immunohistochemistry and ISH +) must have received anti-HER2 therapy, and participants who have not received prior anti-PD-(L)1 or anti-HER2 therapy must have had a contraindication or reasonable reason for no benefit] and have had disease progression.
3. High expression of **CLDN18. 2 was confirmed by pathological examination.

Inclusion Criteria for Phase Ib Cohort B:

1. Histopathologically confirmed unresectable locally advanced or metastatic G/GEJ AC.
2. Disease progression after first-line standard therapy (HER2-overexpressing participants must have received prior anti-HER2 therapy unless contraindicated or justified non-benefit).
3. Confirmed * CLDN18.2-positive by histopathological examination.

Inclusion Criteria for Phase Ib Cohort C:

1. Histopathologically confirmed unresectable locally advanced or metastatic PDAC.
2. Disease progression after at least one prior systemic therapy.

Inclusion criteria for Phase Ib Cohort D:

1. Histopathologically confirmed unresectable locally advanced or metastatic BTC.
2. Disease progression after at least one prior systemic therapy.
3. Confirmed * CLDN18.2-positive by histopathological examination.

Notes:

* CLDN18.2-positive: defined as ≥ 1% of tumor cells with membranous staining of any intensity in tumor tissue by immunohistochemistry, when tested previously, at the study site, or at the central laboratory.

  * High expression of CLDN18. 2: Claudin18.2 immunohistochemical membrane staining intensity ≥ 2 + in ≥ 75% of tumor cells.

    * Moderate to high expression of CLDN18.2: Claudin18.2 immunohistochemical membrane staining intensity ≥ 2 + in ≥ 40% of tumor cells.

      * Specified expression of CLDN18.2: Claudin18.2 immunohistochemical membrane staining intensity 1+/2+/3+ in ≥50% of tumor cells.

Exclusion Criteria:

Exclusion criteria common to Phases Ia and Ib:

1. Is participating in another interventional clinical study other than an observational (non-interventional) clinical study or is in the survival follow-up phase of an interventional study.
2. Has received the last dose of antineoplastic therapy within 4 weeks or 5 half-lives of an antineoplastic therapy (whichever is shorter) prior to the first dose of study drug.
3. Plans to receive other anti-tumor therapy during treatment with the study drug [palliative radiotherapy for symptomatic relief (e.g., pain) that does not affect response assessment is allowed].
4. Has received a strong cytochrome P450 3A4 (CYP3A4) inhibitor within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study drug.
5. Toxicities due to prior therapy that have not recovered to Grade 0 or 1 per NCI CTCAE v5.0 prior to the first dose of study drug (excluding alopecia, asthenia, hyperpigmentation, and other conditions with no safety risk per the judgment of the investigator).
6. Has undergone major surgical procedure (craniotomy, thoracotomy, laparotomy or others per the investigator, excluding needle biopsy) or has unhealed wounds, ulcers, or bone fracture within 4 weeks prior to the first dose of study drug; Or plans to undergo major surgery during the study period; Note: Local surgical treatment of isolated lesions for palliative purposes is acceptable.
7. Has gastric pyloric obstruction and/or persistent recurrent vomiting (≥ 3 episodes in 24 hours).
8. Has a history of gastrointestinal perforation and/or fistula within 6 months that has not resolved surgically prior to the first dose of study drug.
9. Has symptomatic central nervous system metastases. Participants with asymptomatic brain metastases (i.e., no neurological symptoms, no need for glucocorticoid treatment, all brain metastasis ≤ 1. 5 cm) or stable symptoms after treatment of brain metastases must meet all of the following criteria to participate in the study: no metastasis in the midbrain, pons, cerebellum, meninges, medulla oblongata or spinal cord; Stable clinical status for at least 4 weeks with definitive clinical evidence of no new or enlarging brain metastasis and discontinuation of corticosteroids and anticonvulsants for at least 2 weeks prior to the first dose of study drug. Note: lesions of the central nervous system will not be considered as a target lesion
10. Has a history of pneumonitis requiring corticosteroids therapy, or a history of interstitial lung disease, non-infectious pneumonitis, severely impaired lung function or uncontrolled lung disease, such as pulmonary fibrosis, severe radiation pneumonitis, acute lung injury, or suspected of having the above diseases during the screening period.
11. Has uncontrolled medical conditions, such as:
12. Active or clinically uncontrolled serious infection requiring treatment with systemic anti-infectives (antibiotics, antivirals, or antifungals) within 1 week prior to the first dose of study drug, including but not limited to the infection of respiratory tract, urinary system, biliary tract infection, etc.
13. Participants infected with human immunodeficiency virus (HIV) (HIV 1/2 antibody positive).
14. Acute or chronic active hepatitis B (defined as hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody positive (HBcAb) with hepatitis B virus DNA copies ≥ 104 copies/mL or ≥ 2000 IU/mL or above the lower limit of detection) or acute or chronic active hepatitis C [hepatitis C virus antibody (HCVAb) positive with HCV RNA > 103 copies/mL]. Participants whose test results are below the above criteria after receiving antiviral therapy with nucleotides, or participants with positive serology but negative HCV-RNA test result are eligible.
15. Has active pulmonary tuberculosis, is being treated with anti-tuberculosis therapy or having received anti-tuberculosis therapy within 1 year prior to the first dose of study drug.
16. Has active syphilis or latent syphilis requiring treatment.
17. Has symptomatic congestive heart failure (New York Heart Association classification NYHA class II-IV), symptomatic or uncontrolled arrhythmia, QTc interval > 480 ms, or personal or family history of congenital long/short QT syndrome.

    For part 3 1L G/GEJ AC and 1L PDAC cohort, the QTc should be calculated based on the average of triplicate screening ECG (using Appendix 4 Calculation Formula of QTcF)
18. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) by standard treatment.
19. Has one or more arterial thromboembolic event, including myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, etc., within 6 months prior to the first dose of study drug.
20. Has received stent implantation in tracheal or digestive tract.
21. Has symptomatic pleural, ascites, or pericardial effusion requiring intervention (e.g., drainage, peritoneal shunt, or cell-free and concentrated ascites reinfusion therapy [CART]). Asymptomatic participants with a small amount of pleural effusion, ascites or pericardial effusion on imaging are allowed. (Drainage and CART are not allowed within 2 weeks prior to screening assessment).
22. Has esophageal or gastric varices that require immediate intervention (e.g., ligature or sclerotherapy) or are considered to be at high risk for bleeding in the opinion of the investigator or consulting gastroenterologist or hepatologist. Participants with evidence of portal hypertension (including splenomegaly on imaging) or a history of prior variceal bleeding must undergo endoscopic evaluation within 3 months prior to the first dose of study drug.
23. Has one or more life-threatening bleeding event or Grade 3 or 4 gastrointestinal/variceal bleeding requiring blood transfusion, endoscopic or surgical treatment within 3 months prior to the first dose of study drug
24. Has a history of deep vein thrombosis, pulmonary embolism, or any other serious venous thromboembolism within 3 months prior to the first dose of study drug (implantable venous access port or catheter-derived thrombosis, or superficial vein thrombosis is not considered "serious" venous thromboembolism).
25. Has hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh B or more severe cirrhosis.
26. Has complete or incomplete intestinal or bowel obstruction at the time of screening or a history of complete or incomplete intestinal or bowel obstruction within 3 months prior to first dose, or is at risk of intestinal perforation (including but not limited to acute diverticulitis, history of intra-abdominal abscess), or a history of any of the following disease: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection with concurrent chronic diarrhea), Crohn's disease, ulcerative colitis, and chronic diarrhea.
27. Has other acute or chronic disease or laboratory abnormality that may result in increased risk associated with study participation or study drug administration, or interfere with the interpretation of study results, and is considered unfit for this study per the Investigator's judgement.
28. Has a neurological or psychiatric illness or a social situation that affects compliance with study requirements, significantly increases the risk of AE, or affects the participant's ability to provide written ICF.
29. Has a history of other primary malignancies, with the following exceptions:
30. Curatively treated malignancy with no known active disease for ≥ 2 years prior to study enrollment and is at minimal risk of recurrence;
31. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease recurrence;
32. Adequately treated carcinoma in situ with no evidence of disease recurrence.
33. Has a known history of immunodeficiency.
34. Has a history of allogeneic organ transplantation and history of allogeneic hematopoietic stem cell transplantation.
35. Has a history of severe allergic reaction to other monoclonal antibodies and/or hypersensitivity to any of the formulation components of IBI343 or mFOLFOX or Irinotecan or liposomal Irinotecan (For phase 1a part 3 1L G/GEJ AC and 1L PDAC cohort).
36. Female participants who are pregnant or lactating.
37. Has other conditions considered not eligible to participate in this study per the Investigator's judgement.
38. Has known dihydropyrimidine dehydrogenase deficiency (DPD). (NOTE: Screening for DPD deficiency should be conducted per local requirements.)
39. Has known peripheral sensory neuropathy > grade 1 unless the absence of deep tendon reflexes is the sole neurological abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events(AEs), treatment emergent adverse event (TEAEs)，serious adverse events (SAEs) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0.
Dose-limiting Toxicity (DLT) | 21 days after the first dose of IBI343
  DLTs are assessed during the DLT observation period to determine maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).
To determine RP2D of IBI343. | Up to 2 years
  To determine RP2D of IBI343.
ORR assessed by the investigator based on RECIST version 1.1. | Up to 2 years
  ORR assessed by the investigator based on RECIST version 1.1.ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR)
Number of subjects with clinically significant changes in physical examination results | Up to 2 years
  A complete physical examination will include: general appearance, respiratory, cardiovascular, abdomen, skin, head and neck (including ears, eyes, nose, and pharynx), lymph nodes, thyroid, musculoskeletal (including spine and extremities), genital/anal, and neurological assessments, if indicated. Clinically significant abnormal findings at screening will be recorded as medical history or AE based on the investigator's analysis and judgment.
Number of participants with abnormal vital signs | Through study completion, up to 2 years
  Collection of vital signs will include temperature in ℃, measurement tool is physiological parameter
Objective response rate (ORR) | ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR)
  Through study completion, up to 2 years
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Blood routine：RBC, HGB, HCT, WBC, PLT, LYM, ANC
Number of participants with abnormal vital signs | Through study completion, up to 2 years
  Collection of vital signs will include pulse in beats per minute. measurement tool is physiological parameter
Number of participants with abnormal vital signs | Through study completion, up to 2 years
  Collection of vital signs will include respiratory rate in times/min. measurement tool is physiological parameter
Number of participants with abnormal vital signs | Through study completion, up to 2 years
  Collection of vital signs will include blood pressure in kPa. measurement tool is physiological parameter
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Blood biochemistry: TBIL, DBIL, ALT, AST, γ-GGT, ALP, ALB, TP, LDH, Urea or BUN, Cr, Na, K, Cl, Mg, Ca, P, Amylase, Lipase and FBG
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Urinalysis: PH, Specific Gravity, UWBC, UPRO, URBC, UGLU, UBLD
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Coagulation function: APTT, PT, INR, Fbg, D-dimer
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Viral serology test: HBsAg, HBsAb, HBcAb, HBeAg, HBeAb, HBV DNA, HCV antibody, HCV RNA, HIV antibody, Treponema pallidum-specific antibody
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Myocardial injury markers: CK, CK-MB, Troponin I or T, BNP or NT-proBNP
Number of participants with abnormal laboratory tests results | Through study completion, up to 2 years
  Fecal analysis: occult blood (OB)

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Up to 2 years
  PK parameters maximum concentration (Cmax) of IBI343, total antibody, can will be determined.
area under the curve (AUC) | Up to 2 years
  PK parameters area under the curve (AUC) of IBI343, total antibody, exatecan will be determined.
clearance rate (CL) | Up to 2 years
  PK parameters clearance rate of IBI343, total antibody, exatecan will be determined .
half-life (t1/2) | Up to 2 years
  PK parameters half-life (t1/2) of IBI343, total antibody, exatecan will be determined .
Anti-drug antibody(ADA) of IBI343 | Up to 2 years
  The incidence and characterization of ADA of IBI343 will be determined
Objective response rate (ORR) | Through study completion, up to 2 years
  ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR).
time to response (TTR) | Through study completion, up to 2 years
  TTR is defined as the time from the date of first dose of study drug to the date of first documented tumor response (CR/PR).
duration of response (DoR) | Through study completion, up to 2 years
  DoR is defined as the time from the date of first documented tumor response (CR/PR) until PD/death.
disease control rate (DCR) | Through study completion, up to 2 years
  DCR is defined as the proportion of participants with a complete response (CR) or partial response (PR) or stable disease(SD)
progression-free survival (PFS) | Through study completion, up to 2 years
  PFS is defined as the time from the date of first dose of study drug to the date of the first documented progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Through study completion, up to 2 years
  OS is defined as the time from the date of first dose of study drug until the date of death from any cause.
apparent volume of distribution (V) | Up to 2 years
  PK parameters apparent volume of distribution(V) of IBI343, total antibody, exatecan will be determined when appropriate.
Tmax | Up to 2 years
  PK parameters time to maximum concentration of IBI343, total antibody, exatecan will be determined when appropriate.
assess the immunogenicity of IBI343. | Up to 2 years
  The incidence of ADA.
To evaluate the correlation between CLDN18.2 expression level in tumor tissue and anti-tumor activities of IBI343 combination therapy. | Up to 2 years
  Baseline CLDN18.2 expression level and relationship with efficacy.
To evaluate the correlation between CLDN18.2, PD-L1, HER2 expression level in tumor tissue in 1L G/GEJ AC cohort. | Up to 2 years
  Baseline CLDN18.2, PD-L1, HER2 expression level and their correlation in 1L G/GEJ AC cohort.
To determine qualitative metabolic profile of the free payload exatecan in blood or plasma. | Up to 2 years
  For the metabolite profiling cohort only: Relative amounts of exatecan and various other metabolites present in blood or plasma.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (3):
  - NEXT Austin, Austin, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT San Antonio, San Antonio, Texas
- Australia (4):
  - St Vincent Hospital, Darlinghurst, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
- China (32):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Tumor Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital Sun Yat-Sen university, Guangzhou, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangzhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technolog, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Ningxia Medical University General Hospital, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo Medical Center Li Huili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Yang J, Sun Y, Gong J, Yue J, Pan Y, Sun M, Song R, Xiao X, Tazbirkova A, Ruan J, Liu Z, Liu Z, Li Z, Sheng L, Qin Y, Ying J, Yu X, Zhang J, Mou Y, Lu C, Chen P, Li S, Li J, Qu X, Deng T, Du J, Zhou A, Li E, Yuan X, Liang X, Yu W, Morris M, Luo Y, Zhao X, Guo Y, Zhou H, Shen L. CLDN18.2-targeting antibody-drug conjugate IBI343 in advanced gastric or gastroesophageal junction adenocarcinoma: a phase 1 trial. Nat Med. 2025 Sep;31(9):3028-3036. doi: 10.1038/s41591-025-03783-8. Epub 2025 Jul 16. PMID 40670773